CLINICAL TRIAL: NCT02956915
Title: Evaluation of Length of Stay and Predisposing Factors of Late Discharge After Transfemoral Transcatheter Aortic Valve Implantation Using the SAPIEN-3 Prosthesis: A French Multicenter Prospective Observational Trial
Brief Title: Evaluation of Length of Stay After TF-TAVI
Acronym: FAST-TAVI
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/012/HP
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Severe Symptomatic Aortic Stenosis
Keywords: Transcatheter aortic valve implantation; SAPIEN-3 prostheses; Length of stay; Aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with severe symptomatic aortic stenosis: Stable patients with severe symptomatic aortic stenosis undergoing planned Transfemoral Transcatheter aortic valve implantation with the SAPIEN-3 prosthesis will be included. TF-TAVI will be done using a minimalist approach of local anesthesia and conscious sedation.
  Interventions: Procedure: Transfemoral Transcatheter aortic valve implantation

INTERVENTIONS:
Procedure: Transfemoral Transcatheter aortic valve implantation — Transcatheter aortic valve implantation (TAVI): The SAPIEN-3 prosthese are implanted without open heart surgery. The valve delivery system is inserted in the body via the femoral artery.

SUMMARY:
Transcatheter aortic valve implantation (TAVI) has been rapidly adopted worldwide since the first-in-man TAVI performed in 2002. With increasing experience and improvements in valve design, the "minimalist" approach to transfemoral TAVI (using local anesthesia and fluoroscopic guidance) has become an attractive concept, and the technical feasibility of this approach has been well documented.

While earlier data showed prolonged length of stay after TF-TAVI [10.5 ± 8.1 days in the FRANCE 2 registry and 10.2 ± 11.1 days in the PARTNER Cohort A data, the UK TAVI registry (reference) showed a decline in post-TAVI length of stay from 10 days to 8 days over the time period of 2007 to 2012. More contemporary data from other centers has been published showing that 23% of TF-TAVI patients were discharged within 3 days after TAVI. With an increasingly minimalist approach to TF-TAVI, the duration of monitoring required post-procedure remains indeterminate with a lack of formal consensus.

Early discharge (within 3 days of TAVI) is hypothesized to have multiple potential advantages, including reduction in unnecessarily lengthy hospitalization of frail and elderly patients in addition to cost-saving benefits. Rouen University Hospital has previously published a retrospective study on the feasibility and safety of early discharge, in which discharge within 72 hours of uncomplicated TF-TAVI was safe and attained in 36% of our patients. Pre-existing pacemaker and the absence of acute kidney injury were independent predictors of a successful early discharge. Moreover, in a prospective study, Rouen University Hospital recently shown that early discharge afterelective TF-TAVI with SAPIEN-XT/SAPIEN-3 prostheses was attainable in a large proportion of patients (59%) with no evident compromise in safety. Factors associated with failure of early discharge were postprocedural blood transfusion and permanent pacemaker implantation. But currently, there are no guidelines for the length of stay after a TF-TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Stable patients with severe symptomatic aortic stenosis
* Patient undergoing planned TF-TAVI with the SAPIEN-3 prosthesis,
* TF-TAVI using a minimalist approach of local anesthesia and conscious sedation

Exclusion Criteria:

* The use of other (than Edwards SAPIEN-3 or XT) transcatheter aortic valve devices.
* TF-TAVI requiring general anesthesia or surgical cut-down.
* TF-TAVI performed in unstable patients or on an urgent/emergent basis.
* Non-transfemoral routes of valve delivery (eg. transapical, transaortic, etc).
* Discharge back home impossible (including transfer in another hospital)
* Programmed transfer to another hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing an elective TF-TAVI procedure with a SAPIEN-3 prosthesis at participating centers
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of length of stay and reasons for prolonged hospitalization beyond 3 days | 30 days after TF TAVI procedure

SECONDARY OUTCOMES:
Incidence of early discharge/prolonged hospitalization in the overall study population | 30 days after TF TAVI procedure
  Length of stay will be calculated from TAVI procedure (day 0) to discharge
Safety of early discharge | 30 days after TF TAVI procedure
  Combined endpoint of mortality or rehospitalization at 30-days after TF-TAVI procedure
Predictors of early discharge success or failure by multivariate analysis | 30 days after TF TAVI procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hélène ELTCHANINOFF, Pr, Principal Investigator — University Hospital, Rouen
Locations (5):
- France (5):
  - Brest University Hospital, Brest
  - Jacques Cartier Private Hospital, Massy
  - AP-HP Bichat - Claude Bernard Hospital, Paris
  - Rennes University Hospital, Rennes
  - Rouen University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No